CLINICAL TRIAL: NCT00144092
Title: High Dose Chemotherapy and Autologous or Allogeneic Blood Stem Cell Transplantation for Mantle Cell and Relapsed Low Grade Non-hodgkin's Lymphoma
Brief Title: HDCT and Stem Cell Transplantation for Mantle Cell and Relapsed Low Grade Non-hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alberta Health services (Other)
Organization: AHS Cancer Control Alberta (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 147; 15841
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2011-08

CONDITIONS: Low Grade Lymphoma
Keywords: autologous and allogeneic stem cell transplantation; low grade lymphoma; mantle cell
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

INTERVENTIONS:
Procedure: stem cell source

SUMMARY:
Low grade lymphoma patients receive R-ICE reinduction therapy followed by allogeneic stem cell transplanation.

DETAILED DESCRIPTION:
Low grade lymphoma patients receive R-ICE reinduction therapy followed by allogeneic stem cell transplanation if they have an HLA matched sibling, or an autologous transplant if they do not.

ELIGIBILITY:
Inclusion Criteria:

* indolent histology lymphomas after relapse 1 or 2 LVEF > 50% Creatinine < 150 umol/L bilirubin < 30 umol/L wbc >3.5X10^9/L platelets >100X10^9/L other medical condition as controlled

Exclusion Criteria:

* pregnant lactating HIV positive CNS involvement by lymphoma other malignancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2001-05; Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
feasibility
mortality
overall survival
event free survival

CONTACTS AND LOCATIONS:
Overall Officials: Doug Stewart, Principal Investigator — Alberta Cancer Board - TBCC
Locations (1):
- Tom Baker Cancer Centre, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Stewart DA, Duan Q, Carlson L, Russell JA, Bahlis NJ, Duggan P, Hasegawa W, Voralia M. A prospective phase II study of RICE re-induction, then high-dose fludarabine and busulfan, followed by autologous or allogeneic blood stem cell transplantation for indolent b-cell lymphoma. Clin Lymphoma Myeloma Leuk. 2011 Dec;11(6):475-82. doi: 10.1016/j.clml.2011.06.012. Epub 2011 Aug 10. PMID 21831743